CLINICAL TRIAL: NCT01180127
Title: Study of the Impact of a Flavanol Containing Food Product and Exercise on Cognitive Function and Brain Structure
Brief Title: Mars Flavanol Exercise and Cognitive Function Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Mars, Inc. (Industry)
Responsible Party: Principal Investigator, Richard Sloan, Research Scientist, New York State Psychiatric Institute
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 5804
Record Dates: First submitted 2010-05-21; First posted 2010-08-11 (Estimated); Results first posted 2015-01-27 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Cognitive Function
Keywords: flavonol; exercise; dentate gyrus; cerebral blood volume; dentate gyrus CBV
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- exercise, dietary intervention (Active Comparator): aerobic training and flavanol containing food product for 12 weeks
  Interventions: Dietary Supplement: Flavanol containing food product; Behavioral: Aerobic training
- no exercise, dietary intervention (Active Comparator): wait list control plus flavanol containing food product for 12 weeks
  Interventions: Dietary Supplement: Flavanol containing food product; Behavioral: Wait list control
- exercise, food product lacking flavanol (Active Comparator): aerobic training plus food product without flavanol for 12 weeks
  Interventions: Behavioral: Aerobic training; Dietary Supplement: Food product lacking flavanol
- wait list control food additive without flavanol (Placebo Comparator): wait list control plus food product without flavanol for 12 weeks
  Interventions: Dietary Supplement: Food product lacking flavanol; Behavioral: Wait list control

INTERVENTIONS:
Dietary Supplement: Flavanol containing food product — 12 weeks, 2X/day, 20g serving
  Arms: exercise, dietary intervention; no exercise, dietary intervention
Behavioral: Aerobic training — 4X/week, 1 hour/session at 75% maximum HR
  Arms: exercise, dietary intervention; exercise, food product lacking flavanol
Dietary Supplement: Food product lacking flavanol — 20 g serving, 2X/day, food additive lacking flavonol
  Arms: exercise, food product lacking flavanol; wait list control food additive without flavanol
Behavioral: Wait list control — 12 week wait list control condition during which participants abstain from aerobic exercise
  Arms: no exercise, dietary intervention; wait list control food additive without flavanol

SUMMARY:
This is a randomized controlled trial to test the impact of a flavonol containing food product and aerobic exercise on cognitive function and brain structure.

DETAILED DESCRIPTION:
I. Background and Significance A. The epidemiology of cognitive aging. Encompassing multiple cognitive domains, higher order thinking includes memory, language, abstract reasoning, and visuospatial ability. A range of studies have established that memory is a cognitive domain differentially targeted by the normal aging process. With an increase in lifespan and a decrease in co-morbid diseases, aging individuals expect to lead cognitively-challenging lives. Even mild forgetfulness, therefore, is no longer considered 'benign'. Indeed, with the exponential growth of the aging population, and since memory decline will occur in all of us as we age, age-related memory decline has emerged as a major societal problem.

B. The anatomy of cognitive aging. A range of studies in humans, non-human primates and rodents have established that the hippocampal formation, a brain circuit vital for memory, is targeted by the aging process. Age-related hippocampal dysfunction is therefore a major contributor to age-related memory decline.

The hippocampal formation is organized as a circuit, made up of separate but interconnected regions, including the entorhinal cortex, the dentate gyrus, the CA subfields, and the subiculum. Because of hippocampal circuit properties, dysfunction in one subregion will affect the function of neighboring subregions and the hippocampal circuit as a whole. Thus, when confronted with any process that causes the hippocampal circuit to malfunction, pinpointing the subregion that is most effected becomes an important goal.

In the case of age-related memory decline, a range of studies in humans, non-human primates, and rodents, have suggested that normal aging causes hippocampal dysfunction by differentially targeting the dentate gyrus.

C. Imaging cognitive aging. The anatomical organization of the hippocampal circuit and the differential vulnerability of the dentate gyrus to cognitive aging imposes specific requirements on brain imaging techniques. Specifically, an imaging technique must be able to assess the functional integrity of the multiple hippocampal subregions, in particular the dentate gyrus. With this in mind, our lab has been dedicated to optimizing a functional brain imaging approach applicable to both the human and rodent hippocampal formation. We have recently achieved this goal, and have been applying our cross-species imaging capabilities to investigate a range of process that affect hippocampal function.

D. Flavanols, exercise, and cognitive aging. Previous studies have established that physical exercise improved hippocampal function. We have recently exploited our cross-species imaging techniques to show, that within the hippocampal circuit, exercise has a selective effect on dentate gyrus function, in humans and in mice. Independently, a recent study has shown that the flavanol epichatechin improves hippocampal function, and importantly, within the hippocampal circuit, epichatechin was found to differentially target the dentate gyrus. Moreover, this study showed that epichatechin coupled with exercise had its greatest effect on dentate gyrus function.

E. Summary. Starting at around 30 years of age, all of us will begin experiencing the insidious cognitive slide of age-related memory decline. With the expansion of aging, age-related memory decline is swelling to epidemic proportions, and ameliorating age-related memory decline has emerged as major societal goal.

This proposal is designed to test the following hypothesis: That flavanols with or without physical exercise will ameliorate age-related memory decline. This hypothesis is informed by two sets of interleaving findings: First, a range of studies have pinpointed dysfunction in the dentate gyrus as a specific brain region contributing to age-related memory decline; and second, flavanol consumption with or without physical exercise enhances memory performance by improving dentate gyrus function.

In order to experimentally test this hypothesis an imaging technique is required that can assess the functional integrity of the dentate gyrus, techniques that are now available. Importantly, these imaging techniques have been developed so that can they can be applied not only to humans but also to animal models, generating the same 'imaging readout'. Cross-species imaging is particularly important for translational studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-75
2. English-speaking
3. Ambulatory
4. BMI < 32
5. Post-menopausal (women only), no estrogen replacement therapy
6. VO2max < 36 and 33 ml/kg/min for men age 50-59 and 60-69 respectively; < 29 and 27 ml/kg/min for women age 50-59 and 60-75 respectively.
7. Baecke Physical Activity Sports Score ≤ 2
8. Medical clearance to participate in the study (normal serum electrolyte, BUN, creatinine levels, normal blood pressure and resting cardiogram)

Exclusion Criteria:

1. Use of psychotropic medications
2. Current psychiatric disorder
3. Any condition for which aerobic training is counter-indicated
4. Habitual consumers of dietary or herbal supplements, including Gingko, flavonoid, and dietary herbal or plant extracts
5. Lactose Intolerance
6. Individuals who report directly to any of the study investigators
7. Diabetes

Exclusion Criteria (MRI-related)

1. Cardiac Pacemaker
2. Internal Pump
3. Insulin Pump
4. Tattoo eyeliner
5. Wire Sutures
6. Internal Metal Objects
7. Metal Slivers in Eye
8. Prosthesis
9. Hearing Aid Implants
10. Neurostimulator
11. Metal Fragments
12. Brain Aneurysm Clips
13. Vascular Clips
14. Breast Expander
15. Vena Cava Filter
16. Heart Valve
17. Metal Stents
18. Asthma
19. Hay-Fever
20. Sickle Cell Disease
21. Kidney Disease
22. Pregnant

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Small, MD, Principal Investigator — Columbia University

REFERENCES:
- [Background] Pereira AC, Huddleston DE, Brickman AM, Sosunov AA, Hen R, McKhann GM, Sloan R, Gage FH, Brown TR, Small SA. An in vivo correlate of exercise-induced neurogenesis in the adult dentate gyrus. Proc Natl Acad Sci U S A. 2007 Mar 27;104(13):5638-43. doi: 10.1073/pnas.0611721104. Epub 2007 Mar 20. PMID 17374720

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise, Dietary Intervention: aerobic training and flavanol containing food product
  Flavanol containing food product: 12 weeks, 2X/day, 20g serving
  Aerobic training: 4X/week, 1 hour/session at 75% maximum HR
- no Exercise, Dietary Intervention: wait list control plus flavanol containing food product for 12 weeks
  Flavanol containing food product: 12 weeks, 2X/day, 20g serving
  Wait list control: 12 week wait list control condition during which participant abstain from aerobic exercise
- Exercise, Food Additive Lacking Flavanol: aerobic training plus food additive without flavanol
  Aerobic training: 4X/week, 1 hour/session at 75% maximum HR
  Placebo food additive: 20 g serving, 2X/day, food additive lacking flavanol
- Wait List Control Food Additive Without Flavanol: 12 weeks of wait list control status plus food additive without the flavanol containing food product
  Placebo food additive: 20 g serving, 2X/day, food additive lacking flavanol
  Wait list control: 12 week wait list control condition during which participant abstain from aerobic exercise
Period: Overall Study
Arm/Group | Exercise, Dietary Intervention | no Exercise, Dietary Intervention | Exercise, Food Additive Lacking Flavanol | Wait List Control Food Additive Without Flavanol
Started | 10 | 11 | 10 | 10
Completed | 8 | 11 | 9 | 9
Not Completed | 2 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Exercise, Food Additive Lacking Flavonol: aerobic training plus food additive without flavanol
  Aerobic training: 4X/week, 1 hour/session at 75% maximum HR
  Placebo food additive: 20 g serving, 2X/day, food additive lacking flavanol
- Wait List Control Food Additive Without Flavonol: 12 weeks of wait list control status plus food additive without the flavanol containing food product
  Placebo food additive: 20 g serving, 2X/day, food additive lacking flavanol
  Wait list control: 12 week wait list control condition during which participant abstain from aerobic exercise
- Total: Total of all reporting groups
Arm/Group | Exercise, Dietary Intervention | no Exercise, Dietary Intervention | Exercise, Food Additive Lacking Flavonol | Wait List Control Food Additive Without Flavonol | Total
Number analyzed (Participants) | 10 | 11 | 10 | 10 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (4.9) | 57.5 (5.34) | 56.6 (5.56) | 56.6 (3.7) | 57.5 (4.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 7 | 7 | 29
  Male | 2 | 4 | 3 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3 | 4 | 10
  Not Hispanic or Latino | 9 | 9 | 7 | 6 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 2 | 7
  White | 7 | 6 | 6 | 4 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 2 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 10 | 10 | 41

OUTCOME MEASURES:

1. Primary Outcome: CBV-fMRI (Cerebral Blood Volume-functional Magnetic Resonance Imaging)
Description: In steady state conditions, CBV is an indirect measure of basal metabolism in the brain. CBV-fMRI is a technique that generates maps of basal metabolism across different brain regions
Time Frame: Up to 12 weeks after exercise/dietary intervention exposure
Population: One subject in the exercise, food additive lacking flavanol arm, and one subject in the wait list control food additive without flavanol arm had non useable data for this outcome which is why there are only 8 subjects analyzed in those two arms rather than 9.
Measure: Mean (Standard Deviation); unit: percent CBV in a brain region
Arm/Group | Exercise, Dietary Intervention | no Exercise, Dietary Intervention | Exercise, Food Additive Lacking Flavanol | Wait List Control Food Additive Without Flavanol
Number analyzed (Participants) | 8 | 11 | 8 | 8
percent CBV in a brain region
  Baseline | 3.43 (1.43) | 2.55 (0.45) | 2.89 (0.70) | 3.38 (0.52)
  12 weeks | 4.58 (1.66) | 4.48 (1.31) | 2.91 (0.81) | 2.60 (0.59)
Statistical Analysis 1: Comparison: Exercise, Dietary Intervention vs no Exercise, Dietary Intervention vs Exercise, Food Additive Lacking Flavanol vs Wait List Control Food Additive Without Flavanol; Repeated measures ANOVA for the interaction of time (baseline vs 12 week) and flavanol group; Test type: Superiority or Other; p = .0001, Repeated measures ANOVA

2. Primary Outcome: ModBent (Modified Benton Visual Retention Test)
Description: This is an object recognition task. Participants view a complex stimulus, then are asked to select which one of two objects was identical to the studied stimulus. After a series of these matching trials, during the subsequent recognition trials participants are shown serially individual complex objects and asked to indicate whether the object was identical to any of the target stimuli viewed during the matching trials. Their reaction time for correct responses, measured in milliseconds, is the unit of measurement.
Time Frame: Up to 12 weeks after exercise/dietary intervention exposure
Population: One subject in the exercise, dietary intervention and one subject in the no exercise, dietary intervention group had outlying (larger than 3 standard deviation from mean) ModBent values that were deleted and hence those groups have 7 and 10 subjects analyzed rather than 8 and 11 respectively.
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Exercise, Dietary Intervention: aerobic training and flavonol containing food product
  Flavonol containing food product: 12 weeks, 2X/day, 20g serving
  Aerobic training: 4X/week, 1 hour/session at 75% maximum HR
- no Exercise, Dietary Intervention: wait list control plus flavonol containing food product for 12 weeks
  Flavonol containing food product: 12 weeks, 2X/day, 20g serving
  Wait list control: 12 week wait list control condition during which participant abstain from aerobic exercise
- Exercise, Food Additive Lacking Flavonol: aerobic training plus food additive without flavonol
  Aerobic training: 4X/week, 1 hour/session at 75% maximum HR
  Placebo food additive: 20 g serving, 2X/day, food additive lacking flavonol
- Wait List Control Food Additive Without Flavonol: 12 weeks of wait list control status plus food additive without the flavonol containing food product
  Placebo food additive: 20 g serving, 2X/day, food additive lacking flavonol
  Wait list control: 12 week wait list control condition during which participant abstain from aerobic exercise
Arm/Group | Exercise, Dietary Intervention | no Exercise, Dietary Intervention | Exercise, Food Additive Lacking Flavonol | Wait List Control Food Additive Without Flavonol
Number analyzed (Participants) | 7 | 10 | 9 | 9
milliseconds
  Baseline | 1945 (584) | 2296 (1056) | 2291 (515) | 2347 (919)
  12 weeks | 1867 (478) | 2009 (815) | 2560 (1086) | 2794 (1298)
Statistical Analysis 1: Comparison: Exercise, Dietary Intervention vs no Exercise, Dietary Intervention vs Exercise, Food Additive Lacking Flavonol vs Wait List Control Food Additive Without Flavonol; ANCOVA used to test main effect of flavanol; Test type: Superiority or Other; p = 0.038, ANCOVA — The ANCOVA model included a main effect for both flavanol and exercise, so this p-value is for the effect of flavanol on Modbent controlling for baseline Modbent and exercise
Statistical Analysis 2: Comparison: Exercise, Dietary Intervention vs no Exercise, Dietary Intervention vs Exercise, Food Additive Lacking Flavonol vs Wait List Control Food Additive Without Flavonol; ANCOVA used to test main effect of exercise; Test type: Superiority or Other; p = 0.815, ANCOVA — The ANCOVA included both a main effect for flavanol and exercise, so this p-value is for the test of exercise controlling for baseline Modbent and flavanol

3. Secondary Outcome: Modified Rey Auditory Verbal Learning Test
Description: Participants are read a list of words over three learning trials and the subject is asked to free recall as many words as possible after each trial. These 3 trials are followed by 1 learning trial of a distracter list and then a short delayed free recall trial of the initial list. After approximately 60-minutes, subjects are asked to freely recall words from the initial list, then to recall words form the distracter list, and then complete a forced-choice recognition trial. A source memory trial is administered in which subjects are read each presented word and then asked to identify whether they were initially presented during the 3 learning trials or during the distracter trial. Measured as a retention score (ratio) for which the number of words recalled after the short delay is divided by the number of words recalled on the third learning trial.
Time Frame: Up to 12 weeks after exercise/dietary intervention exposure
Population: There were 4 subjects (1 in exercise, dietary intervention; 2 in no exercise, dietary intervention, and 1 in exercise, food additive lacking flavanol) who did not have useable data and are thus not included in analyses.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Exercise, Dietary Intervention | no Exercise, Dietary Intervention | Exercise, Food Additive Lacking Flavanol | Wait List Control Food Additive Without Flavanol
Number analyzed (Participants) | 7 | 9 | 8 | 9
ratio
  Baseline | 0.76 (0.21) | 0.69 (0.19) | 0.80 (0.19) | 0.89 (0.11)
  12 weeks | 0.83 (0.08) | 0.65 (0.25) | 0.76 (0.23) | 0.87 (0.21)
Statistical Analysis 1: Comparison: Exercise, Dietary Intervention vs no Exercise, Dietary Intervention vs Exercise, Food Additive Lacking Flavanol vs Wait List Control Food Additive Without Flavanol; ANCOVA for testing main effect of flavanol; Test type: Superiority or Other; p = 0.853, ANCOVA
Statistical Analysis 2: Comparison: Exercise, Dietary Intervention vs no Exercise, Dietary Intervention vs Exercise, Food Additive Lacking Flavanol vs Wait List Control Food Additive Without Flavanol; ANCOVA for testing main effect of exercise; Test type: Superiority or Other; p = 0.581, ANCOVA

4. Secondary Outcome: VO2max
Description: measured at randomization, i.e., before exposure to the intervention, and then again after completion of the 12-week intervention
Time Frame: Up to 12 weeks after exercise/dietary intervention exposure
Population: One subject in the exercise, dietary intervention and one subject in the exercise, food additive lacking flavanol group had unusable data for this outcome and thus are not included in these analyses.
Measure: Mean (Standard Deviation); unit: mL/(kg·min)
Arm/Group | Exercise, Dietary Intervention | no Exercise, Dietary Intervention | Exercise, Food Additive Lacking Flavanol | Wait List Control Food Additive Without Flavanol
Number analyzed (Participants) | 7 | 11 | 8 | 9
mL/(kg·min)
  Baseline | 25.6 (3.77) | 26.26 (4.62) | 25.1 (4.36) | 23.94 (3.81)
  12 weeks | 27.8 (4.33) | 25.36 (3.66) | 25.98 (6.57) | 25.44 (5.51)
Statistical Analysis 1: Comparison: Exercise, Dietary Intervention vs no Exercise, Dietary Intervention vs Exercise, Food Additive Lacking Flavanol vs Wait List Control Food Additive Without Flavanol; ANCOVA was used to test for an exercise effect; Test type: Superiority or Other; p = 0.237, ANCOVA

ADVERSE EVENTS:
Arm/Group | Exercise, Dietary Intervention | no Exercise, Dietary Intervention | Exercise, Food Additive Lacking Flavonol | Wait List Control Food Additive Without Flavonol
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No